CLINICAL TRIAL: NCT03056352
Title: Metoclopramide for Post-Traumatic Headache. A Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Professor, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-7511
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Metoclopramide; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metoclopramide (Experimental): Metoclopramide 20mg + diphenhydramine 25mg administered intravenously over 15 minutes
  Interventions: Drug: Metoclopramide; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Metoclopramide — Intravenous medication drip
  Other Names: Reglan
Drug: Diphenhydramine — Intravenous medication drip
  Other Names: Benadryl

SUMMARY:
Post-traumatic headache is common. We are determining short and longer-term outcomes among patients treated for post-traumatic headache with IV metoclopramide.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic injury to the head has occurred
* Headache has developed within 7 days of injury to the head
* Headache is not better accounted for by another diagnosis (eg, previous history of migraine or tension-type headache)
* The headache must be rated as moderate or severe in intensity at the time of initial evaluation.
* The plan of the attending emergency physician must include treatment with parenteral metoclopramide.

Exclusion Criteria:

* Patients will be excluded if more than ten days have elapsed since the head trauma, if the headache has already been treated with an anti-dopaminergic medication, or for medication contra-indications including pheochromocytoma, seizure disorder, Parkinson's disease, use of monoamine oxidase inhibitors, and use of anti-rejection transplant medications. Patients will not be excluded for pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Per patient
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide
Started | 21
Completed | 20
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Metoclopramide
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Headache Relief
Description: Sustained headache relief is defined as achieving a headache level of "mild" or "none" within two hours and maintaining a level of "mild" or "none" for 48 hours. Patient self-evaluated pain level is solicited every half hour for two hours in the Emergency Department and then by telephone 48 hours after medication administration.
Time Frame: 2 hours thru 48 hours after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide
Number analyzed (Participants) | 20
Participants | 12

2. Secondary Outcome: Post Concussion Symptoms Assessed by Post-concussive Symptom Scale
Description: The post-concussive symptom scale is a questionnaire administered verbally. The post-concussive symptom ranges from 0 to 132. 0= no post-concussive symptoms. 132= severe post-concussive symptoms.
Time Frame: 7 days
Population: 2 patients were lost to followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metoclopramide
Number analyzed (Participants) | 19
units on a scale | 11.4 (21.4)

3. Secondary Outcome: Number of Participants Satisfied With Medication; Assessed by Self-evaluation
Description: Satisfaction is measured by a positive response to the question "Would you want to receive the same medication during a subsequent visit for post-traumatic headache?"
Time Frame: 48 hours after treatment
Population: 2 patients did not provide an answer to this question
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide
Number analyzed (Participants) | 19
Participants | 16

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected every two hours while in the Emergency Department and then by telephone 48 hours after discharge
Arm/Group | Metoclopramide
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide (N=21)
Drowsiness (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03056352/Prot_SAP_000.pdf